CLINICAL TRIAL: NCT02404740
Title: Continuous Noninvasive Estimation of Intracranial Pressure to Assess Ventriculoperitoneal Shunt Malfunction in Patients With Hydrocephalus
Brief Title: Noninvasive Intracranial Pressure and Hydrocephalus Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1995
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Hydrocephalus
Keywords: VP shunted; Normal intracranial pathology; patients
MeSH Terms: conditions — Hydrocephalus | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- VP shunt functioning: No intervention, just a physiological category--patients with VP shunts that are functioning normally.
  Interventions: Device: Pulse oximetry
- VP shunt malfunctioning: No intervention, just a physiological category--patients with VP shunts that are malfunctioning.
  Interventions: Device: Pulse oximetry
- No known intracranial pathology: No intervention, just a physiological category--patients without VP shunts that have no known intracranial pathology.
  Interventions: Device: Pulse oximetry

INTERVENTIONS:
Device: Pulse oximetry — Pulse oximetry

SUMMARY:
Using a pulse oximeter, we have developed an algorithm that estimates intracranial pressure (ICP) based on patients who have had traumatic brain injuries. Patients with hydrocephalus are typically treated with a shunt in order to reduce ICP. At times the shunt can malfunction. We believe that our algorithm will help identify when a hydrocephalus patient's shunt has malfunctioned.

DETAILED DESCRIPTION:
A malfunctioning ventriculoperitoneal (VP) shunt will typically cause a rise in intracranial pressure, which can be difficult to identify without costly imaging. Novel, state-of-the art machine learning techniques can be leveraged to develop an algorithm that noninvasively estimates intracranial pressure. The resulting algorithm will accurately determine the presence or absence of ventriculoperitoneal shunt malfunction in patients with hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 31 days - 35 years
2. Patients seen at Children's Hospital Colorado Neurosurgery clinic, Emergency Department or on an inpatient service
3. Either hydrocephalus patients with a VP shunt in place (with or without suspicion of VP shunt malfunction), or patients with no known intracranial pathology.

Exclusion Criteria:

1. Pregnant patients
2. Incarcerated patients
3. Patients who object at any time to participating in the study.

Ages: 31 Days to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: VP shunted patient, Normal intracranial pathology patient
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2015-02; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The presence or absence of ventriculoperitoneal shunt malfunction in patients with hydrocephalus | baseline
  The algorithm development

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — Childrens Hospital Colorado

IPD SHARING:
Plan to Share IPD: No